CLINICAL TRIAL: NCT03849651
Title: TCRαβ-depleted Progenitor Cell Graft With Additional Memory T-cell DLI, Plus Selected Use of Blinatumomab, in Naive T-cell Depleted Haploidentical Donor Hematopoietc Cell Transplantation for Hematologic Malignancies
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAP2HCT; NCI-2019-00338 (Registry Identifier: NCI)
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Acute Lymphoblastic Leukemia (ALL); Acute Myeloid Leukemia (AML); Myelodysplastic Syndromes (MDS); NK-Cell Leukemia; Hodgkin Lymphoma; Non Hodgkin Lymphoma (NHL); Juvenile Myelomonocytic Leukemia (JMML); Chronic Myeloid Leukemia (CML)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Large Granular Lymphocytic; Hodgkin Disease; Lymphoma, Non-Hodgkin; Leukemia, Myelomonocytic, Juvenile; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Thiotepa; Melphalan; Granulocyte Colony-Stimulating Factor; Filgrastim; Mesna; thymoglobulin; blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Transplant participants (Experimental): Participants receive a conditioning regimen of ATG (rabbit),Cyclophosphamide 60 mg/kg intravenous once daily, mesna, fludarabine, thiotepa, melphalan, followed by HPC,A Infusion(TCRα/β+ and CD19+ depleted),HPC, A infusion (if needed to achieve goal CD34+ cell dose.CD45RA-depleted DLI will be given at least two weeks after engraftment. Blinatumomab will be given at least one week post-DLI, and only to patients with CD19+ malignancies. G-csf 5mcg/kg subcutaneous or intravenous daily until ANC >2000 for 2 consecutive days.
  Cells for infusion are prepared using the CliniMACS system.
  Interventions: Drug: Cyclophosphamide; Biological: Fludarabine; Drug: Thiotepa; Drug: Melphalan; Biological: G-csf; Drug: Mesna; Device: CliniMACS; Biological: ATG (rabbit); Drug: Blinatumomab; Biological: TCRα/β+; Biological: CD19+; Biological: CD45RA-depleted DLI

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide is a nitrogen mustard derivative. It acts as an alkylating agent that causes cross-linking of DNA strands by binding with nucleic acids and other intracellular structures, thus interfering with the normal function of DNA.
  intravenously (IV) once daily (QD) on day -9
  Other Names: Cytoxan
Biological: Fludarabine — Fludarabine phosphate is a synthetic purine nucleoside analog. It acts by inhibiting DNA polymerase, ribonucleotide reductase and DNA primase by competing with the physiologic substrate, deoxyadenosine triphosphate, resulting in inhibition of DNA synthesis.
  fludarabine phosphate IV QD on days -8 to -4
  Other Names: Fludara
Drug: Thiotepa — Thiotepa is a cell-cycle nonspecific polyfunctional alkylating agent.
  Other Names: Thioplex
Drug: Melphalan — Melphalan, a derivative of nitrogen mustard, is a bifunctional alkylating agent. Melphalan is active against tumor cells that are actively dividing or at rest.
  melphalan IV QD on days -2 to -1
  Other Names: Alkeran
Biological: G-csf — G-csf (granulocytic colony stimulating factor), is a biosynthetic hematopoietic agent that is made using recombinant DNA technology in cultures of Escherichia coli. G-CSF stimulates production, maturation and activation of neutrophils. In addition, endogenous G-CSF enhances certain functions of mature neutrophils, including phagocytosis, chemotaxis and antibody--dependent cellular cytotoxicity.
  Other Names: Neupogen; Filgrastim
Drug: Mesna — Mesna is a synthetic sulfhydryl (thiol) compound. Mesna contains free sulfhydryl groups that interact chemically with urotoxic metabolites of oxaza-phosphorine derivatives such as cyclophosphamide and ifosfamide. Following glomerular filtration, mesna disulfide is rapidly reduced in the renal tubules back to mesna, the active form of the drug.
  Other Names: Mesnex
Device: CliniMACS — Cells for infusion are prepared using the CliniMACS
  Other Names: CliniMACS Prodigy
Biological: ATG (rabbit) — Anti-thymocyte globulin is a purified, pasteurized, gamma immune globulin, obtained by immunization of rabbits with human thymocytes.
  rabbit anti-thymocyte globulin IV daily over 6 hours on days -5 to -3,
  Other Names: Thymoglobulin
Drug: Blinatumomab — Blinatumomab is a bispecific CD19-directed CD3 T-cell engager that mediates formation of a synapse between T cells and the CD19+ target cell, resulting in lysis of that CD19+ cell.Blinatumomab will be given to patients with a history of CD19+ malignancy as determined by St. Jude hematopathologist review of current and historical specimens and reports.
  blinatumomab IV for 28 days beginning at least 1 week post-DLI
  Other Names: Blincyto
Biological: TCRα/β+ — IV on day 0 and may receive an additional dose on day 1
Biological: CD19+ — IV on day 0 and may receive an additional dose on day 1
Biological: CD45RA-depleted DLI — infusion IV

SUMMARY:
Patients less than or equal to 21 years old with high-risk hematologic malignancies who would likely benefit from allogeneic hematopoietic cell transplantation (HCT). Patients with a suitable HLA matched sibling or unrelated donor identified will be eligible for participation ONLY if the donor is not available in the necessary time.

The purpose of the study is to learn more about the effects (good and bad) of transplanting blood cells donated by a family member, and that have been modified in a laboratory to remove the type of T cells known to cause graft-vs.-host disease, to children and young adults with a high risk cancer that is in remission but is at high risk of relapse. This study will give donor cells that have been TCRαβ-depleted. The TCR (T-cell receptor) is a molecule that is found only on T cells. These T-cell receptors are made up of two proteins that are linked together. About 95% of all T-cells have a TCR that is composed of an alpha protein linked to a beta protein, and these will be removed. This leaves only the T cells that have a TCR made up of a gamma protein linked to a delta protein. This donor cell infusion will be followed by an additional infusion of donor memory cells (CD45RA-depleted) after donor cell engraftment.

This study will be testing the safety and effects of the chemotherapy and the donor blood cell infusions on the transplant recipient's disease and overall survival.

DETAILED DESCRIPTION:
In this study, participants with high-risk hematologic malignancies undergoing hematopoietic cell transplantation (HCT), who lack an available suitable human leukocyte antigen (HLA) matched related/sibling donor (MSD) or matched unrelated donor (MUD), will receive a TCRαβ-depleted haploidentical donor HCT with additional memory cell DLI. One course of blinatumomab will be empirically added for patients with CD19+ malignancy.

Primary Objectives

* Determine the maximum effective dose for prophylactic CD45RA-depleted DLI when given in the early post-engraftment period.
* Assess the efficacy of TCRαβ-depleted progenitor cell graft with additional memory T-cell DLI, plus selected use of blinatumomab, in haploidentical donor hematopoietic cell transplantation for hematologic malignancies as measured by 1 year EFS (events = relapse, death)

Secondary Objectives

* Assess the safety and feasibility of the addition of blinatumomab in the early post- engraftment period in patients with CD19+ malignancy
* Estimate the incidence of neutrophil and platelet engraftment, malignant relapse,event-free survival per disease subgroups (e.g. ALL vs AML), and overall survival at one-year post-transplantation.
* Estimate incidence and severity of acute and chronic (GVHD).
* Estimate the rate of transplant related mortality (TRM) in the first 100 days after transplantation.
* To measure and describe the pharmacokinetics of rabbit ATG in HCT recipients on this study.

Exploratory Objectives

* Record immune reconstitution parameters, including chimerism analysis, quantitative lymphocyte subsets, T cell receptor excision circle (TREC) analysis, V-beta spectratyping, and lymphocyte phenotype and function.
* Describe the use of additional CD45RA-depleted DLI for recipients who have severe viral infections, disease recurrence or progression, or poor immune reconstitution. Assess and record efficacy of CD45RA-depleted DLI for these conditions, and all adverse events that are related to CD45RA-depleted DLI.

Blinatumomab will be given to patients with a history of CD19+ malignancy as determined by St. Jude hematopathologist review of current and historical specimens and reports. Blinatumomab dosing will begin no sooner than 1 week after CD45RA-depleted DLI and no later than Day +90. There must be no acute GVHD or it must be quiescent. ALT must be less than 5x ULN, bili less than or equal to 1.5x ULN, and creatinine less than or equal to 1.5x ULN.

If more than one family member donor is suitable, then donor selection will be based on several factors including: degree of KIR mismatching, donor-recipient matching of CMV serology, donor-recipient red blood cell compatibility, degree of HLA matching, size of the potential donor, previous use as a donor, presence of donor-specific antibody, and overall health and availability of the potential donor.

A G-CSF mobilized peripheral blood progenitor cell product (identified as HPC,A) is the preferred progenitor cell graft source. Our desired target goal will be 5 x 10^6 CD34+ cells/kg. This number of cells will be necessary to provide an adequate graft, following the various ex vivo manipulations, for prompt reconstitution. More than one collection may be needed to achieve this goal. Donors will undergo a standard hematopoietic progenitor cell mobilization regimen consisting of 5 days of GSF given subcutaneously at 10 micrograms/kilogram. The graft will be collected by leukapheresis on day 5 (and 6 if needed) of G-CSF. The HPC product will typically be collected and infused fresh, however there may be patients or logistical situations that require the HPC product to be collected early, processed, and stored frozen.

ELIGIBILITY:
Inclusion Criteria for Transplant Recipient

* Age less than or equal to 21 years.
* Does not have a suitable HLA-matched sibling donor (MSD) or volunteer 10/10 HLA-matched unrelated donor (MUD) available in the necessary time for progenitor cell donation.
* Has a suitable single haplotype matched (≥ 3 of 6) family member donor.

High risk hematologic malignancy. High risk ALL in CR1. Examples include, but not limited to: t(9;22) with persistent or recurrent transcript, hypodiploid cytogenetics, MRD >1% at the end of induction, M2 or greater marrow at the end of induction, recurrent or rising MRD after induction, Infants with MLL fusion or t(4;11), relapse after prior CART therapy.

ALL in High risk CR2. Examples include, but not limited to t(9;22), BM relapse <36 mo CR1 or <6mo after completion of therapy, any T-ALL, very early (< 6mo CR1) isolated CNS relapse, late BM relapse with poor response to standard reinduction therapy(e.g. MRD positive or recurrence after two blocks), relapse after prior CART therapy.

ALL in CR3 or subsequent.

AML in high risk CR1 (diagnosis of AML includes myeloid sarcoma). Examples include but not limited to: preceding MDS or MDS-related AML, FAB M0, FAB M6, FAB M7 with high risk genetics such as ML not t(1;22), MRD > 0.1% after two cycles of induction, MRD > 1% after one cycle of induction, FLT3-ITD in combination with NUP98-NSD1 fusion or WT1 mutation, any high risk cytogenetics such as: DEK-NUP214 [t(6;9)], KAT6A-CREBBP [t(8;16)], RUNX1-CBFA2T3 [t(16;21)], -7, -5, 5q-, KMT2A-MLLT10 [t(6;11)], KMT2A-MLLT4 [t(10;11)], inv(3)(q21q26.2), CBFA2T3-GLIS2 [inv(16)(p13.3q24.3)], NUP98-KDM5A [t(11;12)(p15;p13)], ETV6-HLXB [t(7;12)(q36;p13)], NUP98-HOXA9 [t(7;11)(p15.4;p15)], NUP98-NSD1.

AML in CR2 or subsequent.

* Therapy related AML, with prior malignancy in CR > 12mo
* MDS, primary or secondary
* NK cell, biphenotypic, or undifferentiated leukemia in CR1 or subsequent.
* CML in accelerated phase, or in chronic phase with persistent molecular positivity or intolerance to tyrosine kinase inhibitor.
* Hodgkin lymphoma in CR2 or subsequent after failure of prior autologous HCT, or unable to mobilize progenitor cells for autologous HCT.
* Non-Hodgkin lymphoma in CR2 or subsequent after failure of prior autologous HCT, or unable to mobilize progenitor cells for autologous HCT.
* JMML
* If prior CNS leukemia, it must be treated and in CNS CR
* Does not have any other active malignancy other than the one for which this HCT is indicated.
* No prior allogeneic HCT, and no autologous HCT within the previous 12 months.

Patient must fulfill pre-transplant organ function criteria:

* Left ventricular ejection fraction > 40%, or shortening fraction ≥ 25%.
* Creatinine clearance (CrCl) or glomerular filtration rate (GFR) ≥ 50 ml/min/1.73m2.
* Forced vital capacity (FVC) ≥ 50% of predicted value; or pulse oximetry ≥ 92% on room air if patient is unable to perform pulmonary function testing.
* Karnofsky or Lansky (age-dependent) performance score ≥ 50 (See APPENDIX A).
* Bilirubin ≤ 3 times the upper limit of normal for age.
* Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) ≤ 5 times the upper limit of normal for age.
* Not pregnant. If female with child bearing potential, must be confirmed by negative serum or urine pregnancy test within 14 days prior to enrollment.
* Not breast feeding
* Does not have current uncontrolled bacterial, fungal, or viral infection.

Inclusion Criteria for Haploidentical Donor

* At least single haplotype matched (≥ 3 of 6) family member
* At least 18 years of age.
* HIV negative.
* Not pregnant as confirmed by negative serum or urine pregnancy test within 14 days prior to enrollment (if female).
* Not breast feeding.

Regarding donation eligibility, is identified as either:

* Completed the process of donor eligibility determination as outlined in 21 CFR 1271 and agency guidance; OR
* Does not meet 21 CFR 1271 eligibility requirements, but has a declaration of urgent medical need completed by the principal investigator or physician sub-investigator per 21 CFR 1271.

Exclusion Criteria:

-

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-01-31 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2025-08-07 (Estimated)

PRIMARY OUTCOMES:
Maximum effective dose for prophylactic CD45RA-depleted DLI | 90 days after the transplant date of the last enrolled patient.
  Description: A maximum effective dose of CD45RA-depleted DLI is defined as the maximum value of doses that satisfy the proportion of patients with their memory T cell count measured at week 4 post-DLI more than 300/uL is more than 50% and the toxicity of grade 3-4 aGVHD is less than 20%.
One-year Event Free Survival (EFS) after completion of the protocol | One year after the transplant date of the last enrolled patient
  Proportion of patients who are alive and relapse free one year after the date of transplant. (Events=relapse, death)

SECONDARY OUTCOMES:
The number of patients experiencing Blinatumomab permanent discontinuation due to toxicity | 120 days after transplant date of the last enrolled patient
  If the drug is held for more than 2 weeks due to toxicity, it will be permanently discontinued
The estimate of cumulative incidence of relapse | One year after the transplant date of the last enrolled patient
  The cumulative incidence of relapse will be estimated using Kalbfleisch-Prentice method. Death is the competing risk event. The Kaplan-Meier estimates of Overall Survival (OS) and Event Free Survival (EFS) along with their standard errors will be calculated. OS is defined as time from transplantation to death or last follow-up, whichever comes first. EFS is defined as time from transplantation to events including relapse, graft failure, death due to any cause and last follow-up, whichever comes first. The participants are alive at the time of analysis without events will be censored.
The cumulative incidence of acute and chronic Graft-Versus-Host Disease (GVHD) | One year after the transplant date of the last enrolled patient
  The cumulative incidence of acute and chronic (GVHD) will be estimated using Kalbfleisch-Prentice method. Death is the competing risk event. The severity of acute GVHD and chronic GVHD will be described.
The cumulative incidence of transplant related mortality | 100 days after the transplant date of the last enrolled patient
  The cumulative incidence of transplant related mortality will be estimated using Kalbfleisch-Prentice method. Death before day 100 of other reasons are the competing risk events.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Triplett, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols